CLINICAL TRIAL: NCT05650580
Title: A Phase I Clinical Study to Characterize Safety, Tolerability, and Pharmacokinetics of TR115 in Patients With Relapsed / Refractory Non-Hodgkin's Lymphoma or Advanced Solid Tumors
Brief Title: TR115 in Patients With Relapsed / Refractory Non-Hodgkin's Lymphoma or Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tarapeutics Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TR115-CN-PI-01
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Non-Hodgkin's Lymphoma, Relapsed; Non-Hodgkin's Lymphoma Refractory; Advanced Solid Tumor
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose Escalation and Expansion (Experimental): Participants with relapsed/Refractory Non-Hodgkin's Lymphoma or Advanced solid tumor will receive TR115 at escalating and expansion dose levels.
  Interventions: Drug: TR115

INTERVENTIONS:
Drug: TR115 — TR115 is supplied as tablet with dosage strength of 100mg. TR115 tablet will be administered orally on a continuous twice daily (BID) schedule and a treatment cycle is defined as 28 days for the purposes of scheduling procedures and evaluations. TR115 tablets will be given until there appears evidence of progressive disease , intolerable toxicity, or the subject discontinues from the study treatment for other reasons. Proposed daily dose (BID): 100mg, 200mg, 400mg, 800mg, 1200mg, 1600mg. It is possible for additional and/or intermediate dose levels to be added during the course of the study. Cohorts may be added at any dose level below the Maximum Tolerated Dose (MTD) in order to better understand safety, Pharmacokinetic (PK) or Pharmacodynamic (PD).

SUMMARY:
A phase 1 dose escalation and expanded cohort study of TR115 in the treatment of adult patients with relapsed/refractory non-hodgkin's lymphoma or advanced solid tumors.

DETAILED DESCRIPTION:
This is a open-label, dose escalation and expansion, accelerated titration combined 3+3 design, phase 1 study, to evaluate the safety and tolerability, and to determine the Recommeded Phase II Dose (RP2D) of TR115 when administered bid in patients with non-hodgkin's lymphoma or advanced solid tumors. During the dose escalation phase, Up to 6 cohorts of 1-6 0r 3-6 patients each will be treated in the study.

Patients will receive study treatment until criteria for study termination are met. A safety Follow-up Visit will conducted 30 days (±7 days) after the last dose of treatment. Patients who discontinue study treatment for reasons other than disease progression will have post-treatment follow-up for disease assessment until start of new anticancer treatment, lost to follow-up, death, or until the sponsor stops the study, whichever comes first.

After finishing the dose escalation phase, a dose extension phase will be initiated with additional patients included in order to further evaluate the tolerability, pharmacokinetics, and efficacy at the recommended dose that have been evaluated in the dose escalation phase.

Adverse events will be assessed using the NCI Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0.

Tumor response will be assessed by computed tomography (CT) and/or magnetic resonance imaging (MRI) scan using Lugano 2014/RECIST 1.1 criteria, assessed by the investigator.

ELIGIBILITY:
Key Inclusion Criteria:

* fully understand the procedures of the clinical study and participate voluntarily with signed and dated written informed consent form, comply with the requirements of the study protocol.
* males and/or females at least 18 years old when signing the informed consent form.
* tumor type criteria:

  1. relapsed/refractory histologically or cytologically documented non-hodgkin's lymphoma must have received at least 1 prior systemic therapies, including but not limited as below: Follicular Lymphoma (FL), Diffuse Large B-cell Lymphoma (DLBCL), Peripheral T-cell lymphoma-Not Otherwise Specified (PTCL-NOS), Angioimmunoblastic T-cell Lymphoma (AITL), Anaplastic Large Cell Lymphoma (ALCL).
  2. histologically or cytologically confirmed patients with advanced malignant solid tumors, eligible patients must have failed standard treatment, no standard treatment, or not suitable for standard treatment at this stage as determined by the investigator.
* eastern cooperative oncology group performance status (ECOG) ≤2 at screening.
* life expectancy of at least 3 months.
* acceptable organ function: absolute neutrophil count (ANC)≥1.0×109/L (note: growth factor supports within 14 days of the first dose); platelet count (PLT)≥90×109/L （note: PLT≥70 × 109/L for patients with Non-Hodgkin Lymphoma (NHL) and ≥50 × 109/L allowed in patients with bone marrow infiltration. no blood product transfusion is allowed within 14 days of the first dose); hemoglobin (Hb) ≥90g/L (note: Hb ≥80g/L for patients with NHL and ≥70g/L in patients with bone marrow infiltration. no blood product transfusion is allowed within 14 days of the first dose); International Normalized Ratio (INR) or Prothrombin Time (PT)≤1.5×Upper limit of normal value (ULN), Activated Partial Thromboplastin Time (APTT)≤1.5×ULN ；Total bilirubin (TBIL)≤1.5×ULN, Aspartate Amino Tranferase (AST) and Alanine Transaminase (ALT)≤2.5×ULN (note: ≤ 5 × ULN if there is liver involvement); Creatinine (Cr) ≤1.5×ULN or Creatinine Clearance (CCr) ≥50 ml/min (calculated by Cockcroft-Gault formula).
* fertile male and female must agree to use medically approved contraceptives during the study and within 6 months after the last dose of the study.

Key Exclusion Criteria:

* known or suspected allergies to any of the investigational drug compositon.
* medical history and surgical history excluded according to the protocol.
* any previous medical treatment history exclude from the protocol.
* abnormal laboratory results exclude from the protocol.
* pregnant and lactating women (currently breast-feeding or less than six months after delivery although not breast-feeding).
* subjects may not be able to complete the study due to poor compliance or other reasons, or unsuitable for the study by the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-04-23 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events and serious adverse events | from the first dose to within 30 days after the last dose
  frequency, duration and severity of adverse events and serious adverse events evaluated by NCI CTCAE 5.0
dose limited toxicities | within 31 days after the first dose
  incidence of dose limited toxicities
maximum tolerated dose | Throughout the study for approximately 2 years
  evaluated by safety review committee
recommedded phase 2 dose | Throughout the study for approximately 2 years
  evaluated by safety review committee

SECONDARY OUTCOMES:
AUClast | within 31 days after the first dose
  characterize the pharmacokinetic profile of TR115
AUCinf | within 31 days after the first dose
  characterize the pharmacokinetic profile of TR115
Cmax | within 31 days after the first dose
  characterize the pharmacokinetic profile of TR115
Tmax | within 31 days after the first dose
  characterize the pharmacokinetic profile of TR115
CL/F | within 31 days after the first dose
  characterize the pharmacokinetic profile of TR115
Vz/F | within 31 days after the first dose
  characterize the pharmacokinetic profile of TR115
Terminal half-life (T1/2) | within 31 days after the first dose
  characterize the pharmacokinetic profile of TR115

OTHER OUTCOMES:
ORR | Throughout the study for approximately 2 years
  efficacy-overall response rate
PFS | Throughout the study for approximately 2 years
  efficacy-progression free survival
DOR | Throughout the study for approximately 2 years
  efficacy-duration of response
CBR | Throughout the study for approximately 2 years
  efficacy--clinical benefit rate

CONTACTS AND LOCATIONS:
Overall Officials: Jie Jin, MD, PhD, Principal Investigator — Zhejiang University
Locations (1):
- The first affiliated hospital, Zhejiang university school of medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No